CLINICAL TRIAL: NCT03658694
Title: Repetitive Transcranial Magnetic Stimulation of the Precentral-gyrus in the Relief of Fibromyalgia Pain: an International Multicenter Controlled Adaptative Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation of Relief of Fibromyalgia Pain
Acronym: TMSFFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, Pain Center of Department of Neurology, University of Sao Paulo
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RGDCA03
Record Dates: First submitted 2018-09-03; First posted 2018-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is an adaptive sequential trial of FM patients. In stage 1 patients were randomly allocated into two parallel arms (conventional rTMS, sham) using adaptive methodology. In stage 2, after the end of the first trial, patients will be allocated to two arms (conventional rTMS, patterned rTMS). Both stages will be conducted in a sequential methodology where an interim analysis will take place and indicate whether will take place trial is positive and of the scientific board agrees open its start.
  Recruitment time will be extended by 12 months due to dropouts related to the Covid-19 pandemic. We have had dropouts due to some patients who developed Covid-19 and also due to patients who were afraid of becoming infected during hospital visits. Those patients who dropped out of the study due to the pandemic will be excluded from the main analysis and will be analyzed as a secondary outcome.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Conventional rTMS - study 1 (Experimental): In study 1 patients were randomly allocated to receive conventional repetitive transcranial magnetic stimulation (10Hz).
  Interventions: Procedure: Conventional rTMS - study 1
- Sham rTMS - study 1 (Experimental): In study 1 patients were randomly allocated to receive sham repetitive transcranial magnetic stimulation.
  Interventions: Procedure: Sham rTMS - study 1
- Conventional rTMS - study 2 (Experimental): In study 2, after the end of the first trial will be allocated to receive conventional of repetitive transcranial magnetic stimulation (10Hz).
  Interventions: Procedure: Conventional rTMS - study 2
- Patterned rTMS - study 2 (Experimental): In study 2, after the end of the first trial will be allocated to receive patterned of repetitive transcranial magnetic stimulation (Theta-burst).
  Interventions: Procedure: Patterned rTMS - stage 2

INTERVENTIONS:
Procedure: Conventional rTMS - study 1 — Patients will be undergoing to 10Hz transcranial magnetic stimulation session
  Arms: Conventional rTMS - study 1
Procedure: Sham rTMS - study 1 — Patients will be undergoing to sham transcranial magnetic stimulation session
  Arms: Sham rTMS - study 1
Procedure: Conventional rTMS - study 2 — Patients will be undergoing to 10Hz transcranial magnetic stimulation session
  Arms: Conventional rTMS - study 2
Procedure: Patterned rTMS - stage 2 — Patients will be undergoing to theta-burst transcranial magnetic stimulation session
  Arms: Patterned rTMS - study 2

SUMMARY:
There are currently several points concerning rTMS for pain relief that have a huge impact in the practical application of rTMS in clinical practice, but which have not been approached by previous studies. Also, an even more important issue is the frequency of the sessions in each treatment protocol. The idea of performing stimulation in chronic pain patients on a consecutive daily basis for long-term treatments seem unrealistic and potentially costly. However, it has been reported in animals, healthy subjects and FM patients that the analgesic effects of rTMS can outlast the stimulation session for several minutes and even days. This has led to the proposal that pain treatment with rTMS could be performed in consecutive daily induction sessions, followed by spaced (weekly, fortnightly and even monthly) maintenance sessions. This approach is similar to what is performed routinely in patients with major depression treated by rTMS to the dorsolateral prefrontal cortex, and has successfully been tested in FM patients in a single- center study. Should this approach prove effective in larger prospective multicentric studies, rTMS could enter the armamentarium of non-invasive, non- pharmacological, low-adverse event therapeutic options to relieve fibromyalgia- related pain and associate symptoms. Hence, our aim is to conduct a multicentric international clinical trial on the influence of rTMS in the control of pain in a consecutive adaptive trial design where conventional rTMS (10Hz) and patterned rTMS (theta-burst) will be studied. Stimulations will be performed in a clinical practice-friendly approach, where daily maintenance sessions will be followed by weekly, and fortnightly stimulation sessions. There have been very scarce adaptive trials in the pain and non-invasive stimulation fields. This methodological approach allows for the use of lower number of patients in consecutive trials and, among other qualities, it allows for the imputation of data from the first trial into the second one, thus decreasing the duration of the studies and the number of participants.

DETAILED DESCRIPTION:
There are currently several points concerning rTMS for pain relief that have a huge impact in the practical application of rTMS in clinical practice, but which have not been approached by previous studies. One of them refers to dosing of the treatment. rTMS sessions have been proposed to comprise from 1000 to 3000 pulses of stimulation in each session, which means that treatment sessions may last from 7 to 20 minutes. While there are positive studies reporting different numbers of pulses, the actual stimulation protocol chosen may impact not only the efficacy of the treatment, but also the duration of the stimulation session, the time patients stay at the health-care facility, and, thus, cost and compliance to treatment. Also, an even more important issue is the frequency of the sessions in each treatment protocol. The idea of performing stimulation in chronic pain patients on a consecutive daily basis for long-term treatments seem unrealistic and potentially costly. However, it has been reported in animals, healthy subjects and FM patients that the analgesic effects of rTMS can outlast the stimulation session for several minutes and even days. This has led to the proposal that pain treatment with rTMS could be performed in consecutive daily induction sessions, followed by spaced (weekly, fortnightly and even monthly) maintenance sessions. This approach is similar to what is performed routinely in patients with major depression treated by rTMS to the dorsolateral prefrontal cortex, and has successfully been tested in FM patients in a single- center study. Should this approach prove effective in larger prospective multicentric studies, rTMS could enter the armamentarium of non-invasive, non- pharmacological, low-adverse event therapeutic options to relieve fibromyalgia- related pain and associate symptoms. Hence, our aim is to conduct a multicentric international clinical trial on the influence of rTMS in the control of pain in a consecutive adaptive trial design where conventional rTMS and patterned rTMS will be studied. Stimulations will be performed in a clinical practice-friendly approach, where daily maintenance sessions will be followed by weekly, and fortnightly stimulation sessions. There have been very scarce adaptive trials in the pain and non-invasive stimulation fields. This methodological approach allows for the use of lower number of patients in consecutive trials and, among other qualities, it allows for the imputation of data from the first trial into the second one, thus decreasing the duration of the studies and the number of participants. Similarly, this technical approach allows for pre-planned interim analyses to be performed during data collection, allowing for the sample size to be readjusted during the trial, and, more importantly, allowing for trial termination due to futility or due to achievement of the primary endpoint before the end of the original preplanned data collection period, with lower risk of bias. Here, the adaptive approach will allow one not only to compare conventional rTMS (10Hz) to sham stimulation, but also, on second consecutive study, it will provide the first head-to-head study on rTMS to date comparing the analgesic effects of conventional (10Hz) and patterned (theta-burst) rTMS .

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with diagnosis fibromyalgia according to the ACR 2016 criteria (patient satisfies modified 2016 fibromyalgia criteria if the following 3 conditions are met: 1) widespread pain index (WPI) ≥ 7 and symptom severity scale (SSS) score 5 OR WPI of 4-6 and SSS score ≥ 9. 2) Generalized pain, defined as pain in at least 4 of 5 regions, must be present. Jaw, chest, and abdominal pain are not included in generalized pain definition. 3) Symptoms have been generally present for at least 3 months. 4) A diagnosis of fibromyalgia is valid irrespective of other diagnoses. A diagnosis of fibromyalgia does not exclude the presence of other clinically important illnesses).
2. Age ≥18 years;
3. Be able to understand study protocol and give signed, written informed consent
4. Not under opioids
5. VAS score ≥ 40/100 mm;

Exclusion Criteria:

1. Known abuse of alcohol or illicit drugs
2. Known psychiatric conditions
3. Contraindications to rTMS (42) (Head trauma or concussion, metal implants in the skull, pregnancy, cardiac pacemaker, medication infusion devices, previous troubles with TMS or MRI);
4. Not being under chronic contraceptive use (intrauterine dispositive or oral contraceptive)
5. Other medical conditions demand hospitalization;
6. Participation in other clinical studies at the same time

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Analgesic effects of motor cortex stimulation | 8th week of treatment
  Percentage of responders based on the reduction of ≥50% in pain intensity (numerical rating scale 0-10) at the end of the study compared to baseline.

SECONDARY OUTCOMES:
Global impression of change | 8th and 16th weeks of treatment
  Assess % of very much and much improved
Pain intensity | At the end of the induction period (10th day) and 16th week
  Measured by VAS (0 no pain -10 worst pain)
Mood | 8th week of treatment
  Assess mood by hospital anxiety and depression scale
Impact of fibromyalgia daily | 8th and 16th week of treatment
  Assess by fibromyalgia impact questionnaire
Interference in daily activites | 8th week of treatment
  Measured by brief pain inventory
Medication use | 8th week of treatment
  Measured by Brief Pain Inventory
Phenotypical markers of analgesic response | 8th and 16th week of treatment
  Assessment of phenotypical markers of analgesic response
Adverse events | 8th and 16th week of treatment
  Assess of adverse events by standardized questionnaire'

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ciampi de Andrade, MD, PhD, Principal Investigator — Pain Center, Department of Neurology, University of Sao Paulo, Sao Paulo, Brazil
Locations (6):
- Brazil (4):
  - Universidade Federal de Pernambuco, Recife, Pernambuco
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC/FMUSP), São Paulo, São Paulo
  - Federal University of ABC, São Bernardo do Campo
  - Ambulatório de Fisioterapia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Centre d'Evaluation et de Traitement de la Douleur Hôpital Ambroise Paré, Paris, France
- Department of Neuromodulation Osaka University, Osaka, Japan

REFERENCES:
- [Derived] Lins CC, Fonseca AS, Martins PN, Oliveira JCB, Fernandes AM, Baptista AF, Kubota GT, da Silva VA, Teixeira MJ, de Andrade DC. Investigation of predictors of pain relief with high-frequency repetitive motor cortex transcranial magnetic stimulation among people with fibromyalgia. Neurophysiol Clin. 2025 Nov;55(6):103109. doi: 10.1016/j.neucli.2025.103109. Epub 2025 Oct 4. PMID 41046849